CLINICAL TRIAL: NCT06806735
Title: Quantification of Hypertrophic Scar Tissue or Keloid Using a 3D-Camera
Brief Title: Measuring the Volumes of Hypertrophic Scars and Keloids, Two Specific Kind of Scars, Over Different Points in Time in Patients Who Have Undergone Surgery and Evaluate 3D-cameras As a Possible Measuring and Documenting Tool Including Volumetry
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01147
Record Dates: First submitted 2025-01-21; First posted 2025-02-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Keloid Scar Following Surgery; Scars, Hypertrophic; Scar Keloid
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: 3D-Pictures — 3D-Pictures will be taken of hypertrophic scars and keloids to document them.

SUMMARY:
Measuring the volumes of hypertrophic scars and keloids, two specific kind of scars, over different points in time in patients who have undergone surgery and evaluate 3D-cameras as a possible measuring and documenting tool including volumetry.

DETAILED DESCRIPTION:
The objective of this study is to utilize a 3D camera to measure the volumes of hypertrophic scars and keloids in patients at specified time points. The time points for measurement include day 0, as well as 3, 6, and 12 months. The 3D camera will be evaluated for their efficacy in measuring and documenting the volumes of the scars. This evaluation will include volumetry, which is the measurement of the three-dimensional space occupied by an object.

ELIGIBILITY:
Inclusion Criteria:

* All patients with hypertrophic scars or keloids, written consent to participate in the study, minimum age of 18 years.

Exclusion Criteria:

* Absence of written consent, unwillingness to contribute data, inability to understand the study protocol.
* lack of hypertrophic scars or keloid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertrophic scars or keloids of the University Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Measurability | Day 0, Month 3, 6 and 12
  The objective of this study is to determine the feasibility of utilizing 3D cameras to accurately measure hypertrophic scars and keloids. The primary outcome of this study is the measurement of the volumes of hypertrophic scars in cubic millimeters (equivalent to milliliters) over a period of one year. This will allow for an evaluation of the accuracy of 3D photography and for the observation of any potential changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsspital Zürich, Zurich, Canton of Zurich, Switzerland